CLINICAL TRIAL: NCT02099669
Title: Red Blood Cell Transfusion Thresholds and QOL in MDS (EnhanceRBC): a Pilot, Feasibility Study
Brief Title: Red Blood Cell Transfusion Thresholds and QOL in MDS
Acronym: EnhanceRBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Juravinski Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCCMDS-005
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Myelodysplastic Syndromes (MDS); Quality of Life; Red Blood Cell (RBC) Transfusions
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal transfusion strategy (Experimental): Intervention: Red Blood Cell transfusions. Transfuse pRBC at a higher threshold- maintain Hb level between 110 and 120 g/L: to achieve this, 2 units of pRBCs are transfused when Hb level is < 105 g/L and 1 unit of RBCs when Hb level is 105-110 g/L.
  Transfusions administered more frequently.
  Interventions: Other: Red Blood Cell Transfusions
- Restrictive transfusion strategy (Active Comparator): Intervention: Red Blood Cell transfusions. Transfuse pRBC at standard of care thresholds- maintain Hb level between 85 and 100 g/L: to achieve this, 2 units of packed red blood cells (pRBCs) will be transfused when the Hb level is < 80 g/L and 1 unit of pRBCs when Hb level is 80-85 g/L: standard administration
  Interventions: Other: Red Blood Cell Transfusions

INTERVENTIONS:
Other: Red Blood Cell Transfusions

SUMMARY:
Myelodysplastic syndromes (MDS) are bone marrow malignancies characterized by poor bone marrow function that may progress to acute myeloid leukemia. Many patients become red blood cell transfusion-dependent. Transfusion dependence is associated with inferior quality of life (QOL). However, the relationship between the degree of anemia and QOL is less clear. A commonly used transfusion strategy is to target the hemoglobin (Hb) in the range of 80-90 g/L (normal hemoglobin > 120-130g/L). The question is: would a higher hemoglobin target lead to improvement in QOL despite the negative impact transfusion dependence may have on QOL (due to associated time commitments, expense, transfusion reactions etc). Several groups have prospectively shown that targeting hemoglobin levels of greater than 120 g/L (with hematopoietic growth factors (HGFs) and/or blood transfusions) or incremental increases of 15-20 g/L (with HGFs alone) were associated with improved QOL. The investigators MDS program has been conducting prospective assessments of QOL since 2007 in all registered and consented patients using a variety of validated questionnaires. Preliminary analysis (in 236 patients) revealed that, compared with an age-matched healthy general population, MDS patients have inferior QOL. Transfusion dependence and anemia were independently predictive of poor functioning, fatigue and decreased health utility. Furthermore, a hemoglobin level of ≥100 g/L seemed to be the key threshold for improvement in function and symptom scores. The investigators hypothesize that the target hemoglobins in transfusion dependent MDS patients are too low and this may account for their inferior quality of life. Our goal is to compare the effect on QOL of a restrictive strategy (which is the current standard of care), with a liberal transfusion strategy in a large randomized controlled trial of transfusion dependent MDS outpatients. Before embarking on such an endeavor, the investigators must first prove feasibility in a smaller pilot randomized controlled trial.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are bone marrow malignancies characterized by poor bone marrow function that may progress to acute myeloid leukemia. Many patients become red blood cell transfusion-dependent. Transfusion dependence is associated with inferior quality of life (QOL). However, the relationship between the degree of anemia and QOL is less clear. A commonly used transfusion strategy is to target the hemoglobin (Hb) in the range of 80-90 g/L (normal hemoglobin > 120-130g/L). The question is: would a higher hemoglobin target lead to improvement in QOL despite the negative impact transfusion dependence may have on QOL (due to associated time commitments, expense, transfusion reactions etc). Several groups have prospectively shown that targeting hemoglobin levels of greater than 120 g/L (with hematopoietic growth factors (HGFs) and/or blood transfusions) or incremental increases of 15-20 g/L (with HGFs alone) were associated with improved QOL. The investigators MDS program has been conducting prospective assessments of QOL since 2007 in all registered and consented patients using a variety of validated questionnaires. Preliminary analysis (in 236 patients) revealed that, compared with an age-matched healthy general population, MDS patients have inferior QOL. Transfusion dependence and anemia were independently predictive of poor functioning, fatigue and decreased health utility. Furthermore, a hemoglobin level of ≥100 g/L seemed to be the key threshold for improvement in function and symptom scores. The investigators hypothesize that the target hemoglobins in transfusion dependent MDS patients are too low and this may account for their inferior quality of life. Our goal is to compare the effect on QOL of a restrictive strategy (which is the current standard of care), with a liberal transfusion strategy in a large randomized controlled trial of transfusion dependent MDS outpatients. Before embarking on such an endeavor, the investigators must first prove feasibility in a smaller pilot randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients with MDS ≥18 years of age
* Transfusion dependent: at least 1 transfusion per month in the last 8 weeks
* Hb <100g/L pre transfusion
* Life expectancy > 6 months

Exclusion Criteria:

* Unstable cardiac disease (Canadian Cardiovascular Society (CCS) III/IV angina or New York Heart Association (NYHA) III/IV congestive heart failure) requiring the transfusion target range to remain >85-100 g/L at all times
* ECOG ≥3
* Patients with red cell antibodies against high frequency antigens or multiple antibodies (would potentially delay finding blood)
* Patients on ESA's or disease modifying agents (like azacitidine) for their MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Percentage compliance of q2weekly hemoglobins | 3 months
  The percentage compliance of q2weekly hemoglobins being within or above the target range of the RBC transfusion threshold assigned (after the 4 week run-in at study start as defined above). We will consider this study feasible and worthy of future development into a larger randomized trial (powered for QOL difference) if compliance is ≥70%. A compliance rate of 50-70%, would not exclude going forward with such an RCT but only after careful discussion and statistical planning

SECONDARY OUTCOMES:
Measures of feasibility | 3 months
  * Number of patients ineligible due to screen failure
  * Enrolment rates defined by the number of enrolled patients/month
  * Percentage compliance with QOL questionnaire completion at least 3 serial times
  * Other logistical issues related to protocol implementation, recruitment rates, randomization implementation strategy, data collection, patient tolerability of study schedule
Quality of life | 3 months
  • The magnitude of change in physical functioning, fatigue, dyspnea and global health scores on the EORTC QLQ-C30, calculated health utility on the EQ-5D and fatigue score on FACT-F comparing the 2 RBC transfusion thresholds above.
Adverse events | 3 months
  * The rate of transfusion reactions (as defined by TTISS (Transfusion Transmitted Injuries Surveillance System by Public Health Agency of Canada))
  * Rate of adverse events such as cardiac events and thromboembolic events as per NCI CTCAE version 4.0 criteria
Alloimmunization rates | 3 months
  Rate of alloimmunization to significant blood group antigens
Hemosiderosis | 3 months
  • The impact on transfusion associated hemosiderosis rates and burdens (as measured by changes in ferritin levels and iron chelating medications)
Overall utilization of blood | 3 months
  How many units of blood are required to maintain the hemoglobin threshold chosen
Time commitment | 3 months
  • The overall time commitment per group, measured as the time spent in transfusion medicine clinic

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre/Odette Cancer Centre
Locations (3):
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto
  - Sunnybrook Health Sciences Centre/Odette Cancer Centre, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836